CLINICAL TRIAL: NCT00931372
Title: Restoration of First Phase Insulin Release in Subjects With Type 2 Diabetes Mellitus With Subcutaneous Injection of 20 µg AVE0010 in a Double-blind, Randomized, Placebo-controlled, Two-way Cross Over Intravenous Glucose Challenge Study.
Brief Title: Lixisenatide for Restoration of Insulin Release in Subjects With Diabetes Mellitus Type 2
Acronym: RESTORE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Profil GmbH, Neuss, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY10433; EudraCT:2008-003242-28
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin release; Diabetes mellitus type 2; GLP-1 agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: AVE0010/Placebo (Experimental): Period 1: lixisenatide 20 µg in 200 µL, one single dose
  Period 2: placebo 200 µL, one single dose
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Placebo
- Sequence 2: Placebo/AVE0010 (Experimental): Period 1: placebo 200 µL, one single dose
  Period 2: lixisenatide 20 µg in 200 µL, one single dose
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Placebo

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Solution for subcutaneous injection 100 µg/mL
Drug: Placebo — Subcutaneous injection

SUMMARY:
The objective of this study is to test whether Lixisenatide (AVE0010) restores first phase and improves second phase insulin response in subjects with diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with type 2 diabetes mellitus on diet and exercise with/without metformin
* HbA1c>=6,0 % and <=8,5 % at screening
* BMI 25 to 35 kg/m²
* 155>=BP systolic >=90 mmHg
* 100>=BP diastolic>=45 mmHg

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Area under the insulin secretion curve | within 10 minutes after I.V. glucose challenge

SECONDARY OUTCOMES:
Area under the insulin secretion curve | within 10 to 120 minutes after I.V. glucose challenge

CONTACTS AND LOCATIONS:
Overall Officials: Christoph KAPITZA, MD, Principal Investigator — Profil GmbH, Neuss, Germany
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany